CLINICAL TRIAL: NCT01312428
Title: A Prospective Clinical Evaluation of Acetabular Cup Placement in Total Hip Replacements Utilizing a Pelvic Alignment Level (PAL) Instrument
Brief Title: Pelvic Alignment Level (PAL) Instrument Evaluation
Acronym: PAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lagging enrollment
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2015-02

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic Alignment Level (PAL) (Other): Pelvic Alignment Level Instrument Used
  Interventions: Device: Pelvic Alignment Level (PAL) Instrument
- No Pelvic Alignment Level (PAL) (Other): No Pelvic Alignment Level Instrument Used
  Interventions: Device: No Pelvic Alignment Level (PAL) Instrument

INTERVENTIONS:
Device: Pelvic Alignment Level (PAL) Instrument — Pelvic Alignment Level Instrument Used
  Arms: Pelvic Alignment Level (PAL)
Device: No Pelvic Alignment Level (PAL) Instrument — No Pelvic Alignment Level Instrument Used
  Arms: No Pelvic Alignment Level (PAL)

SUMMARY:
The study is conducted to evaluate the performance of the Pelvic Alignment Level (PAL) instrument in achieving desired acetabular position, desired leg length and offset after Total Hip Replacement (THR) reconstruction.

DETAILED DESCRIPTION:
Total hip replacement (THR) has been a sucessful treatment for cases of degenerative joint diseases. However, post operative complications such as dislocations, osteolysis, component wear and migration are still a concern. It has been noted in the scientific literature that precise acetabular cup position helps reduce such post operative complications. The Pelvic Alignment Level (PAL) offers this solution by assessing pelvic motion and optimizing implant position without the need for intra-operative fluoroscopy or a large capital expenditure. The focus of this study is to evaluate the clinical outcomes (acetabular cup placement, femoral offset, and leg length) of using the PAL instrument to those without using PAL instrument during total hip replacement. This will be a prospective, post market, randomized multi-center clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed an IRB approved, evaluation specific Informed Patient Consent Form.
* Patient is a male or non-pregnant female age 18 years or older at time of enrollment.
* Patient clinically qualifies for total hip arthroplastic surgery, based on physical examination and medical history.
* Patient must have a diagnosis of: osteoarthritis, traumatic arthritis, avascular necrosis, slipped capital epiphysis, pelvic fracture, failed fracture fixation or rheumatoid arthritis.

Exclusion Criteria:

* Patient's anatomy precludes a cup placement of 45° inclination and 20° anteversion.
* Patient has an active infection within the affected hip joint.
* Patient is a prisoner.
* Patient has plans to relocate to another geographic area before the completion of the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L. Malkani, MD, Study Chair — Healthcare Center for Advanced Medicine
Locations (1):
- Healthcare Center for Advanced Medicine, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PAL (Pelvic Alignment Level): The cases randomized into the "PAL Group" will have total hip replacement surgery performed utilizing the PAL instrument.
  Pelvic Alignment Level (PAL) Instrument: Total hip replacement surgery will be performed utilizing the PAL Instrument.
- No PAL (No Pelvic Alignment Level): The cases randomized into the "No PAL Group" will have total hip replacement surgery performed without the use of the PAL instrument. This group will serve as the control group.
  Total Hip Replacement: Total hip replacement surgery will be performed without utilizing the PAL Instrument.
Period: Overall Study
Arm/Group | PAL (Pelvic Alignment Level) | No PAL (No Pelvic Alignment Level)
Started | 3 | 4
Completed | 0 | 0
Not Completed | 3 | 4
Not completed — Study Termination | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- PAL (Pelvic Alignment Level): The cases randomized into the PAL group will have total hip replacement surgery performed utilizing the PAL instrument.
  Pelvic Alignment Level (PAL) Instrument: Total hip replacement surgery will be performed utilizing the PAL Instrument.
- No PAL (No Pelvic Alignment Level): The cases randomized into the no PAL group will have total hip replacement surgery performed without the use of the PAL instrument. This group will serve as the control group.
  Total Hip Replacement: Total hip replacement surgery will be performed without utilizing the PAL Instrument.
- Total: Total of all reporting groups
Arm/Group | PAL (Pelvic Alignment Level) | No PAL (No Pelvic Alignment Level) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12.9) | 65.9 (4.1) | 65.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Surgical Accuracy in Placing Acetabular Components at a Target of 45° Inclination and 20° Anteversion While Using the PAL Compared to Surgeries Without Using the PAL Instrument.
Time Frame: 6 week follow-up
Population: The study was terminated early, therefore, primary or secondary measures were not assessed.
Arm/Group | PAL (Pelvic Alignment Level) | No PAL (No Pelvic Alignment Level)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Evaluate the Surgical Success of Achieving Preoperative Targets for Leg Length and Femoral Offset, or be Able to Document Changes to Pre-operative Leg Length and Offset, Using the PAL Compared to Surgeries Without Using the PAL Instrument.
Time Frame: 6 week follow-up
Population: The study was terminated early, therefore, primary or secondary measures were not assessed.
Arm/Group | PAL (Pelvic Alignment Level) | No PAL (No Pelvic Alignment Level)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Industry Standard Adverse Event (AE) terms (e.g. MedDRA) were not used for AE data collection. Specific AE terms were not used for all AEs collected.
Arm/Group | PAL (Pelvic Alignment Level) | No PAL (No Pelvic Alignment Level)
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAL (Pelvic Alignment Level) (N=3) | No PAL (No Pelvic Alignment Level) (N=4)
Operative Site (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To publish, exhibit or lecture, the manuscript, exhibit or speech must be provided to Stryker at least 60 days prior to submission for publication or presentation. The Investigator must receive consent from Stryker prior to publication, exhibition, or disclosure of scientific and clinical data. This review by Stryker is not intended to curtail distribution of scientific and clinical data, but to identify and edit any company confidential material and/or violations of FDA and FTC regulations.